CLINICAL TRIAL: NCT02929784
Title: Assesing Hemiplegic Shoulder Pain and the Use of tDCS to Treat This Pain
Brief Title: tDCS to Treat Hemiplegic Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Loewenstein Hospital (Other)
Responsible Party: Principal Investigator, Motti Ratmansky, MD, Head of pain unit, Loewenstein Hospital, Loewenstein Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: loe160033ctil
Record Dates: First submitted 2016-10-09; First posted 2016-10-11 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Stroke
Keywords: Hemiplegic Shoulder Pain; transcranial Direct Current Stimulation; Stroke
MeSH Terms: conditions — Stroke | interventions — Methods

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Electrode positioning will be determined according to the EEG 10-20 international system for EEG electrode placement: Affected hemisphere anodal stimulation of the hand area of the primary motor cortex (C3/C4), Intensity of 2 mA (milliampere) for duration of 20 minutes. A total of 10 sessions: 5 sessions a week for 2 weeks.
  Interventions: Device: Intervention
- Sham (Sham Comparator): The stimulator will be turned on for only a very short duration of time (msec) no meaningful stimulation is believed to be administered in such a way.
  Interventions: Device: Sham
- no HSP (No Intervention): Patients hospitalized in the Loewenstein department of neurologic rehabilitation after first clinical stroke who do not have hemiplegic shoulder pain.

INTERVENTIONS:
Device: Intervention — Device: neuroConn_CE_DC-STIMULATOR. Anodal stimulation to affected hemisphere.
  Arms: Intervention
Device: Sham — no meaningful stimulation will be given.
  Arms: Sham

SUMMARY:
The purpose of the study is to investigate the possibility of treating Hemiplegic Shoulder Pain (HSP) using transcranial direct current stimulation (tDCS) in patients following stroke.

The secondary aims are to see if this treatment affects motor function of the upper limb, to asses the different types of HSP and whether there is any correlation to the location and extent of the stroke.

DETAILED DESCRIPTION:
Hemiplegic Shoulder Pain (HSP) is a common entity following stroke. It's prevalence varies between studies, probably because it includes many etiologies and there is no one way of diagnosis.

HSP delays rehabilitation, elongates hospitalization time and reduces quality of life.

Currently there is no one reccomended treatment for HSP. Weak transcranial direct current stimulation (tDCS) induces persisting excitability changes in the human motor cortex. this effect depends on the stimulation polarity and is specific to the site of stimulation. Interacting with cortical activity, by means of cortical stimulation, can improve the rehabilitation potential of neurologic patients. In this respect, preliminary evidence suggests that cortical stimulation may play a role in treating aphasia, unilateral neglect, and chronic pain disorders.

In this tDCS study the investigator uses one anode and one cathode electrode placed over the scalp to modulate a particular area of the central nervous system (CNS). The stimulation is administered via the neuroConn DC.Stimulator. The DC-STIMULATOR is a micro-processor-controlled constant current source. The DCSTIMULATOR is a CE-certified medical device for conducting non-invasive transcranial direct current stimulation (tDCS) on people.Electrode positioning is determined according to the International EEG 10-20 System.

ELIGIBILITY:
Inclusion Criteria:

* Patients hospitalized in the department of neurologic rehabilitation of Loewenstein Rehabilitation Center after first clinical stroke.
* Able to understand and comply with basic instructions
* Signed an informed consent form
* Hebrew speaking

Exclusion Criteria:

* Shoulder pain predating the stroke
* Epilepsy

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2020-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
Change in VAS (Visual Ananlof Scale) for pain assessment | 1 month
  using an validated score 0 (lowest) to 10 (highest)

SECONDARY OUTCOMES:
Change in Fugl-Meyer assessment | 1 month
  The Fugl-Meyer Assessment is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia.Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 226.

CONTACTS AND LOCATIONS:
Overall Officials: Motti Ratmansky, Principal Investigator — Loewenstein Rehabilition Center